CLINICAL TRIAL: NCT04567199
Title: Retrospective Analysis of the Influence of Cytosorb on Catecholamine Reduction and Mortality in SIRS and Sepsis
Brief Title: Influence of Cytosorb on Amount of Catecholamine and Mortality in Sepsis
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1124/2018
Record Dates: First submitted 2020-09-09; First posted 2020-09-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-09

CONDITIONS: Sepsis; Septic Shock; Cytokine Storm; Cytokine Release Syndrome; Catecholamine
MeSH Terms: conditions — Sepsis; Shock, Septic; Cytokine Release Syndrome | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cytosorb recipients: Patients receiving Cytosorb due to septic shock.
  SOFA score, Changes in catecholamine support after CytoSorb initiation Survival to discharge ICU Survival >28d Thromboembolic events
  General data:
  Need of catecholamines Type of extra-corporal treatments Anticoagulation medication Concomitant allogenic blood products Concomitant factor concentrates Bleeding events Vital signs Underlying Disease SAPSII, SAPSIII, SOFA Scores (on 1st day of treatment) Type of Pathogen (gram+, gram-, fungi) Sepsis Multi Organ Failure
  Data records:
  Myoglobin, CK (creatine kinase), CK-MB, Fibrinogen D-dimers, Antithrombin III, Procalcitonin Creatinin, urea, Natrium, Potassium, Bilirubin, GOT (glutamate-oxalacetate transaminase), GPT, GGT (glutamate-pyruvate transaminase), PT (prothrombin time) aPTT (activated partial thromboplastin time) CRP (C reactive protein) Blood count Further parameters if of interest
  Interventions: Other: Observational, retrospective
- Non Cytosorb recipients: Patients not receiving Cytosorb due to septic shock.
  Patients not treated with CytoSorb under suspicion for inflammation, septic shock or SIRS will be searched for same characteristics as the first group.
  These groups will be matched when parameters like epidemiology, infectious parameters, prognostic scores, age, gender amount of catecholamines fit best.
  Parameters as in Group of Cytosorb recipients
  Interventions: Other: Observational, retrospective

INTERVENTIONS:
Other: Observational, retrospective — retrospective analysis of observed results, for both study groups.

SUMMARY:
The aim of this retrospective study was to identify if the enrolled patient might have had a profit of Cytosorb therapy. Primarily the decline in catecholamine therapy under Cytosorb therapy will be investigated. Secondarily the outcome of surviving patients will be evaluated and compared to expected mortality due to sequential organ failure assessment (SOFA). Thirdly the patients deceased under this therapy were compared to the surviving patients.

DETAILED DESCRIPTION:
Severe septic Shock has a high mortality ranging from 30-55% and might lead up to 100% mortality under cardiovascular failure and vasoplegia in the initial phase of severe septic shock . Mostly caused by bacteremia, it can also be triggered by viral or fungal infections. Due to vasodilatation caused by toxins the circulatory system of the patient fails. This will lead to further malfunctions of the patient organs (e.g. renal malfunction, vasodilation, myocardial pump failure and DIG) and will cause multiorgan system failure.

Nowadays there is a symptomatic approach to treat septic shock. Except of giving antibiotics less can be done to improve the patient's condition. Treatment with fluids, catecholamines, mechanical ventilation, renal replacement therapies are all regimen to bridge failed organ systems until normal organ function is restored and starts to improve. It is known that the cytokines and toxins, which are liberated by the breakdown of bacterial cells, maintain the inflammatory response of the body. This process might be overshooting and if not disrupted, the patient will die.

A new approach is to bind this cytokines and toxins in an unspecific physical process to tiny plastic beads, which are arranged in the CytoSorb System as they correlate with severity of mortality in sepsis . This polymer beads allow adsorption and binding of molecules from 5-60 kDa (kilodalton) range. Therefore, Cytokines as IL(interleukin)-1, -6, -8 and -10 can be effectively removed. CytoSorb has to get in contact with patient blood. To use this option of treatment CytoSorb is implemented in a renal replacement system, a heart lung machine, ECMO (extracorporeal membrane oxygenator) or any other extracorporeal pump driven system. By extracorporeal blood purification in septic shock the main goal is to eliminate inflammatory mediators and bacterial toxins. This might attenuate the excessive inflammatory response and could lead to hemodynamic stabilization .

The aim of this retrospective study was to identify if the enrolled patient might have had a profit of Cytosorb therapy. Primarily the decline in catecholamine therapy under Cytosorb therapy will be investigated. Secondarily the outcome of surviving patients will be evaluated and compared to expected mortality due to sequential organ failure assessment (SOFA). Thirdly the patients deceased under this therapy were compared to the surviving patients.

ELIGIBILITY:
Inclusion Criteria:

* No CytoSorb therapy in patient suspected for sepsis or SIRS (systemic inflammatory response syndrome)
* CytoSorb therapy in patient suspected for sepsis or SIRS

Exclusion Criteria:

* no signs of inflammation
* no sepsis
* no SIRS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Due to this relatively new treatment concept there is less data at the moment available. 50 patients treated with CytoSorb, if available, in suspicion of severe septic shock will be examined to collect data on outcome. These patients will be compared to 50 patients not treated with CytoSorb. Overall about 100 patients will be analysed.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Catecholamine rate over time | Begin of Sepsis or Cytosorb [=time 0]; multiple time points (0, 1, 2, 3, 4, 6, 8, 24, 48, 72, 96 hours post timepoint 0
  Change of Catecholamine rate [µg of catecholamine/kilogram of body weight /minute].

SECONDARY OUTCOMES:
Length of stay | Begin of Sepsis until discharge [up to 54 weeks]
  Length of stay in hospital
Overall survival | Begin of Sepsis until discharge [up to 54 weeks]
  Amount of survivors at discharge
28 day survival | Begin of Sepsis and day 28
  Amount of survivors at timepoint day 28 [in % of all patients]

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ströhle, MD, Principal Investigator — Univ.-Klinik für Allgemeine und Chirurgische Intensivmedizin
Locations (1):
- General and Surgical Critical Care Medicine, Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data regarding the patients condition (lab values, catecholamine need, and other parameters)